CLINICAL TRIAL: NCT04713176
Title: A Double-blind, Randomized, Placebo-controlled, Multi-center, Phase III Study to Evaluate the Efficacy and Safety of DW1248 With Remdesivir in Severe COVID-19 Patients
Brief Title: Efficacy and Safety of DWJ1248 With Remdesivir in Severe COVID-19 Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination of study due to sponsor's internal decision
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1248302
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Severe COVID-19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWJ1248 with Remdesivir (Experimental): Camostat mesylate 200 mg, Remdesivir
  Interventions: Drug: DWJ1248 with Remdesivir
- Placebo with Remdesivir (Placebo Comparator): Placebo, Remdesivir
  Interventions: Drug: Placebo with Remdesivir

INTERVENTIONS:
Drug: DWJ1248 with Remdesivir — 1 tablet of DWJ1248 TID(up to 14 days) PO, Remdesivir(up to 5 or 10 days) IV
  Arms: DWJ1248 with Remdesivir
Drug: Placebo with Remdesivir — 1 tablet of placebo TID(up to 14 days) PO, Remdesivir(up to 5 or 10 days) IV
  Arms: Placebo with Remdesivir

SUMMARY:
Efficacy and Safety of DWJ1248 with Remdesivir in Severe COVID-19 Patients

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 19 as of the signed date in written consent
* Subjects with COVID-19 according to RT-PCR test(within 10 days)
* Subjects who need to be hospitalized and injected Remdesivir

Exclusion Criteria:

* Subjects who cannot orally administer the investigational products
* Subjects who requiring mechanical ventilation or ECMO
* Acute Respiratory Distress Syndrome(ARDS), shock, multiple organ dysfunction syndrome
* Subjects who need administration of immunosuppressants
* Subjects who are allergic or sensitive to investigational products or its ingredients
* Crcl < 30 mL/min or eGFR < 30 mL/min/1.73m^2
* AST or ALT >= 5xULN
* Subjects who have been identified with uncontrolled concomitant diseases or conditions, including significant mental illness and social conditions, that may affect compliance with clinical trial procedures according to the determination of the investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Proportion of Subjects with Point 7 or Point 8 in the 8 point ordinal scale during 29 days | Up to 29 days
  Percentage of patients with death(ordinal scale of 8) or ECMO patients(ordinal scale of 7)

SECONDARY OUTCOMES:
Time to recovery | Day 3,5,8,11,15,22,29
Desirable of Outcome Ranking (DOOR) | Day 15,29
  The DOOR is scored by evaluating two items: ordinal scale and serious adverse events.
  DOORs are as follows: 1: Recovery (corresponding to the ordinal scale of 1, 2, or 3); 2: Improvement (reduced by more than 1 score of the ordinal scale compared to baseline) with no serious adverse events; 3: Improvement (reduced by more than 1 score of the ordinal scale compared to baseline) with serious adverse events; 4: No change (no change in the ordinal scale compared to baseline) with no serious adverse events; 5: No change (no change in the ordinal scale compared to baseline) with serious adverse event regardless of causality; 6: Deterioration (increased by more than 1 score of the ordinal scale compared to baseline); 7: Death
Duration of Hospitalization | Day 29
  The duration of hospitalization (days)
Time to death | Day 15,29
  The percent of participants

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Center, Seoul, South Korea